CLINICAL TRIAL: NCT04494867
Title: Core Warming of COVID-19 Patients Undergoing Mechanical Ventilation: a Randomized, Single Center Pilot Study
Brief Title: Core Warming in COVID-19 Patients Undergoing Mechanical Ventilation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sharp HealthCare (Other)
Collaborators: Advanced Cooling Therapy, Inc., d/b/a Attune Medical (Industry)
Responsible Party: Principal Investigator, David Willms, MD, Director, Clinical Care Services, Sharp HealthCare
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: COVID-19 Core Warming
Record Dates: First submitted 2020-07-29; First posted 2020-07-31 (Actual); Results first posted 2023-03-09 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-02

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Core warming (Experimental): Patients receive the Attune Medical Esophageal Heat Transfer Device (EnsoETM) and undergo core warming
  Interventions: Device: Core Warming
- Standard of Care (Active Comparator): Patients receive standard temperature management and treatment
  Interventions: Other: Standard of Care

INTERVENTIONS:
Device: Core Warming — Esophageal heat transfer device will be set to 42°C temperature after initial placement, and maintained at 42°C for the duration of treatment.
  Other Names: EnsoETM
  Arms: Core warming
Other: Standard of Care — Standard temperature management and treatment
  Arms: Standard of Care

SUMMARY:
The purpose of the proposed pilot study is to determine if core warming improves respiratory physiology of mechanically ventilated patients with COVID-19, allowing earlier weaning from ventilation, and greater overall survival.

DETAILED DESCRIPTION:
This is a small scale pilot study to evaluate if core warming improves respiratory physiology of mechanically ventilated patients with COVID-19, allowing earlier weaning from ventilation, and greater overall survival. This prospective, randomized study will include 20 patients diagnosed with COVID-19, and undergoing mechanical ventilation for the treatment of respiratory failure. Patients will be randomized in a 1:1 fashion with 10 patients (Group A) randomized to undergo core warming, and the other 10 patients (Group B) serving as the control group who will not have the ensoETM device used. Patients randomized to Group A will have core warming initiated in the ICU or other clinical environment in which they are being treated after enrollment and provision of informed consent from appropriate surrogate or legally authorized representative.

ELIGIBILITY:
Inclusion Criteria:

* Patients above the age of 18 years old.
* Patients with a diagnosis of COVID-19 on mechanical ventilation.
* Patient maximum baseline temperature (within previous 12 hours) < 38.3°C.
* Patients must have a surrogate or legally authorized representative able to understand and critically review the informed consent form.

Exclusion Criteria:

* Patients without surrogate or legally authorized representative able to provide informed consent.
* Patients with contraindication to core warming using an esophageal core warming device.
* Patients known to be pregnant.
* Patients with <40 kg of body mass.
* Patients with DNR status.
* Patients with acute stroke, post-cardiac arrest, or multiple sclerosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-08-19 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Willms, MD, Principal Investigator — Sharp HealthCare; Ahmed Salem, MD, Principal Investigator — Sharp HealthCare
Locations (1):
- Sharp Memorial Hospital, San Diego, California, United States

REFERENCES:
- [Background] Evans EM, Doctor RJ, Gage BF, Hotchkiss RS, Fuller BM, Drewry AM. The Association of Fever and Antipyretic Medication With Outcomes in Mechanically Ventilated Patients: A Cohort Study. Shock. 2019 Aug;52(2):152-159. doi: 10.1097/SHK.0000000000001368. PMID 31058720
- [Background] Drewry AM, Ablordeppey EA, Murray ET, Dalton CM, Fuller BM, Kollef MH, Hotchkiss RS. Monocyte Function and Clinical Outcomes in Febrile and Afebrile Patients With Severe Sepsis. Shock. 2018 Oct;50(4):381-387. doi: 10.1097/SHK.0000000000001083. PMID 29240644
- [Background] Drewry AM, Ablordeppey EA, Murray ET, Stoll CRT, Izadi SR, Dalton CM, Hardi AC, Fowler SA, Fuller BM, Colditz GA. Antipyretic Therapy in Critically Ill Septic Patients: A Systematic Review and Meta-Analysis. Crit Care Med. 2017 May;45(5):806-813. doi: 10.1097/CCM.0000000000002285. PMID 28221185
- [Background] Drewry AM, Fuller BM, Skrupky LP, Hotchkiss RS. The presence of hypothermia within 24 hours of sepsis diagnosis predicts persistent lymphopenia. Crit Care Med. 2015 Jun;43(6):1165-9. doi: 10.1097/CCM.0000000000000940. PMID 25793436
- [Background] Drewry AM, Fuller BM, Bailey TC, Hotchkiss RS. Body temperature patterns as a predictor of hospital-acquired sepsis in afebrile adult intensive care unit patients: a case-control study. Crit Care. 2013 Sep 12;17(5):R200. doi: 10.1186/cc12894. PMID 24028682
- [Background] Drewry AM, Hotchkiss R, Kulstad E. Response to "Body temperature correlates with mortality in COVID-19 patients". Crit Care. 2020 Jul 24;24(1):460. doi: 10.1186/s13054-020-03186-w. No abstract available. PMID 32709253
- [Derived] Bonfanti NP, Mohr NM, Willms DC, Bedimo RJ, Gundert E, Goff KL, Kulstad EB, Drewry AM. Core Warming of Coronavirus Disease 2019 Patients Undergoing Mechanical Ventilation: A Pilot Study. Ther Hypothermia Temp Manag. 2023 Dec;13(4):225-229. doi: 10.1089/ther.2023.0030. Epub 2023 Aug 2. PMID 37527424

RESULTS

PARTICIPANT FLOW:
Groups:
- Core Warming: Patients assigned to receive the Attune Medical Esophageal Heat Transfer Device (EnsoETM) and undergo core warming
  Core Warming: Esophageal heat transfer device will be set to 42°C temperature after initial placement, and maintained at 42°C for the duration of treatment.
- Standard of Care: Patients assigned to receive standard temperature management and treatment
  Standard of Care: Standard temperature management and treatment
Period: Overall Study
Arm/Group | Core Warming | Standard of Care
Started | 10 | 10
Completed | 7 | 6
Not Completed | 3 | 4

BASELINE CHARACTERISTICS:
Population: Patients who were randomized and received either core warming treatment or standard of care treatment. Does not include patients were randomized and withdrawn from study prior to receiving treatment.
Groups:
- Core Warming: Patients who received the Attune Medical Esophageal Heat Transfer Device (EnsoETM) and undergo core warming
  Core Warming: Esophageal heat transfer device will be set to 42°C temperature after initial placement, and maintained at 42°C for the duration of treatment.
- Standard of Care: Patients who received standard temperature management and treatment
  Standard of Care: Standard temperature management and treatment
- Total: Total of all reporting groups
Arm/Group | Core Warming | Standard of Care | Total
Number analyzed (Participants) | 9 | 10 | 19
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 5 | 6 | 11
  >=65 years | 4 | 4 | 8
Age, Continuous [Median (Standard Deviation); unit: years] | 61.7 (15.1) | 59.4 (10.3) | 60.5 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 3 | 7
  Male | 5 | 7 | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 9 | 10 | 19
Time to Enrollment [Mean (Standard Deviation); unit: days] | 9.4 (13.1) | 9.1 (11.8) | 9.3 (12.1)
Height [Mean (Standard Deviation); unit: meters] | 1.623 (0.104) | 1.687 (0.098) | 1.66 (0.10)
Weight [Mean (Standard Deviation); unit: kilograms] | 94.8 (23.5) | 95.2 (14.2) | 95.1 (18.6)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 35.8 (7.8) | 33.4 (3.4) | 34.5 (5.9)
Tobacco Usage [Count of Participants; unit: Participants] | 1 | 1 | 2
Ethanol Usage [Count of Participants; unit: Participants] | 1 | 3 | 4
Pre-Existing Cardiovascular Condition [Count of Participants; unit: Participants] | 6 | 8 | 14
Pre-Existing Respiratory Condition at Baseline [Count of Participants; unit: Participants] | 6 | 7 | 13
Pre-Existing Hepatic Condition [Count of Participants; unit: Participants] | 2 | 4 | 6
Pre-Existing Gastrointestinal Condition [Count of Participants; unit: Participants] | 1 | 5 | 6
Pre-Existing Genitourinary Condition at Baseline [Count of Participants; unit: Participants] | 3 | 4 | 7
Pre-Existing Endocrine Condition [Count of Participants; unit: Participants] | 8 | 8 | 16
Pre-Existing Hematologic Condition [Count of Participants; unit: Participants] | 5 | 6 | 11
Pre-Existing Musculoskeletal Condition [Count of Participants; unit: Participants] | 6 | 8 | 14
Pre-Existing Neoplastic Condition [Count of Participants; unit: Participants] | 0 | 1 | 1
Pre-Existing Neurologic Condition [Count of Participants; unit: Participants] | 2 | 2 | 4
Pre-Existing Psychiatric Condition [Count of Participants; unit: Participants] | 2 | 1 | 3
Pre-Existing Immunologic Condition [Count of Participants; unit: Participants] | 3 | 5 | 8
Pre-Existing Dermatologic Condition [Count of Participants; unit: Participants] | 0 | 0 | 0
Pre-Existing HEENT Condition [Count of Participants; unit: Participants] | 1 | 1 | 2
Other Pre-Existing Condition [Count of Participants; unit: Participants] | 3 | 3 | 6
Allergies [Count of Participants; unit: Participants] | 0 | 1 | 1
Baseline Cycle Threshold [Mean (Standard Deviation); unit: Cycles] | 31.7 (1.6) | 27.1 (1.45) | 29.1 (4.8)

OUTCOME MEASURES:

1. Primary Outcome: PaO2/FiO2 Ratio
Description: Determine the change in PaO2/FiO2 ratio at 0, 24, 48, and 72 hours after implementation of core warming of ventilated patients, and compare this change to patients undergoing standard care.
Time Frame: 0, 24, 48, and 72 hours after initiation of core warming
Measure: Mean (Standard Error); unit: Ratio
Arm/Group | Core Warming | Standard of Care
Number analyzed (Participants) | 9 | 10
Ratio
  0-hour timepoint | 119.1435 (11.57574) | 164.789 (19.42075)
  24-hour timepoint | 130.0138 (17.01536) | 154.9758 (21.10532)
  48-hour timepoint | 158.2389 (19.43118) | 196.7167 (30.56792)
  72-hour timepoint | 134.3884 (13.41839) | 196.9593 (32.0182)

2. Secondary Outcome: Cycle Threshold at 72-hours
Description: Determine the change cycle threshold after implementation of core warming of ventilated patients, and compare this change to patients undergoing standard care.
Time Frame: 72 hours after initiation of core warming
Measure: Mean (Standard Deviation); unit: Cycles
Arm/Group | Core Warming | Standard of Care
Number analyzed (Participants) | 9 | 10
Cycles | 31.4 (3.2) | 30.8 (6.4)

3. Secondary Outcome: Ventilator-Free Days
Description: Measure the impact of core warming on duration of mechanical ventilation.
Time Frame: Initiation of Core Warming Until Patient Weaned Off Mechanical Ventilation
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Core Warming | Standard of Care
Number analyzed (Participants) | 9 | 10
days | 6.8 (10.2) | 11.9 (12.6)

4. Secondary Outcome: 30-Day Mortality
Description: Determine impact of core warming on patient mortality.
Time Frame: 30 days after initiation of core warming
Measure: Count of Participants; unit: Participants
Arm/Group | Core Warming | Standard of Care
Number analyzed (Participants) | 9 | 10
Participants | 2 | 4

ADVERSE EVENTS:
Time Frame: Until 30 days post randomization or until hospital discharge
Arm/Group | Core Warming | Standard of Care
All-Cause Mortality (participants affected / at risk) | 2/9 | 4/10
Serious Adverse Events (participants affected / at risk) | 1/9 | 2/10
Other Adverse Events (participants affected / at risk) | 9/9 | 9/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Core Warming (N=9) | Standard of Care (N=10)
MSSA Bacteremia (Infections and infestations) | 1 (1) | 0 (0)
Stenotrophomonas maltophilia pneumonia and bacteremia (Infections and infestations) | 0 (0) | 1 (1)
Worsening of bilateral upper/lower extremity weakness (Nervous system disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Core Warming (N=9) | Standard of Care (N=10)
Fever (Infections and infestations) | 0 (0) | 1 (1)
Diabetes mellitus (Endocrine disorders) | 1 (1) | 1 (1)
tachycardia (Cardiac disorders) | 2 (2) | 2 (2)
fungal infection (Infections and infestations) | 0 (0) | 1 (1)
headache (Nervous system disorders) | 0 (0) | 1 (1)
elevated D-dimer (Immune system disorders) | 1 (1) | 2 (2)
delirium (Nervous system disorders) | 0 (0) | 2 (2)
hypertension (Cardiac disorders) | 0 (0) | 1 (1)
hypertriglyceridemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
elevated liver function tests (Hepatobiliary disorders) | 2 (2) | 2 (2)
anemia (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
adrenal insufficiency (Renal and urinary disorders) | 0 (0) | 1 (1)
E. coli pneumonia (Infections and infestations) | 0 (0) | 1 (1)
hypotension (Cardiac disorders) | 0 (0) | 1 (1)
pseudomonas aeruginosa pneumonia (Infections and infestations) | 0 (0) | 1 (1)
tracheobronchitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
E. coli bacteremia (Infections and infestations) | 0 (0) | 1 (1)
hypernatremia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
premature atrial contractions (Cardiac disorders) | 0 (0) | 1 (1)
hepatic steatosis (Hepatobiliary disorders) | 0 (0) | 1 (1)
penile skin yeast infection (Infections and infestations) | 0 (0) | 1 (1)
elevated procalcitonin (Immune system disorders) | 2 (2) | 1 (1)
PTH intact (Endocrine disorders) | 0 (0) | 1 (1)
septic shock (Infections and infestations) | 1 (1) | 1 (1)
supraglottic edema (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
dysphagia (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
stammering (Nervous system disorders) | 0 (0) | 1 (1)
stool positive for occult blood (Gastrointestinal disorders) | 0 (0) | 1 (1)
toxic vacuoles (Immune system disorders) | 0 (0) | 1 (1)
elevated troponin (Cardiac disorders) | 0 (0) | 1 (1)
elevated eosinophils (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
leukocytosis (Immune system disorders) | 2 (2) | 1 (1)
bacterial superinfection (Infections and infestations) | 1 (1) | 0 (0)
azotemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
mild respiratory alkalosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
heparin-induced thrombocytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
possible herpes stomatitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
hyperammonia cholestasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
hyperglycemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
toxic metabolic encephalopathy (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
low phosphorous level (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
femoral DVT (Vascular disorders) | 1 (1) | 0 (0)
Klebsiella pneumonia (Infections and infestations) | 1 (1) | 0 (0)
aortic valve stenosis (Cardiac disorders) | 1 (1) | 0 (0)
head tremor (Nervous system disorders) | 1 (1) | 0 (0)
pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
tracheostomy leak (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
tracheostomy wound infection (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
tracheobronchomalacia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
elevated PTT (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
mastoiditis (Infections and infestations) | 1 (1) | 0 (0)
hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
elevated BUN (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
tinea corpus under pannus (Infections and infestations) | 1 (1) | 0 (0)
anasarca (Vascular disorders) | 1 (1) | 0 (0)
epistaxis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
acute encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
elevated CA-125 tumor marker (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
elevated carcino-embyonic antigen (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
leukopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
sepsis (Infections and infestations) | 1 (1) | 0 (0)
acute tubular necrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
duodenal ulcers (Gastrointestinal disorders) | 1 (1) | 0 (0)
tongue deviation (Nervous system disorders) | 1 (1) | 0 (0)
hypokalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
enterobacter penumonia (Infections and infestations) | 1 (1) | 0 (0)
elevated RDW (Blood and lymphatic system disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-03-02): https://cdn.clinicaltrials.gov/large-docs/67/NCT04494867/Prot_SAP_000.pdf